CLINICAL TRIAL: NCT00913133
Title: Multi-Center Trial of Desirudin for the Prophylaxis of Thrombosis: an Alternative to Heparin-Based Anticoagulation (DESIR-ABLE)
Brief Title: Safety Study of Desirudin, an Anticoagulant for the Prophylaxis of Thrombosis
Acronym: DESIR-ABLE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Canyon Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DES-09-02
Record Dates: First submitted 2009-05-26; First posted 2009-06-04 (Estimated); Results first posted 2013-01-03 (Estimated); Last update posted 2013-01-10 (Estimated); Status verified 2013-01

CONDITIONS: Thrombosis
Keywords: Anticoagulation; Prophylaxis; Desirudin; Direct thrombin inhibitor; Heparin-induced thrombocytopenia
MeSH Terms: conditions — Thrombosis | interventions — desirudin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Desirudin (Experimental): desirudin 15 mg twice daily for a minimum of 5 days
  Interventions: Drug: Desirudin

INTERVENTIONS:
Drug: Desirudin — Desirudin SC 15mg q12h
  Other Names: Iprivask

SUMMARY:
The objective of this trial is to demonstrate the clinical utility of fixed-dose SC Desirudin for the prophylaxis of thrombosis as an alternative to heparin-based anticoagulation.

DETAILED DESCRIPTION:
Hospitalized patients who require DVT prophylaxis and who are not good candidates for heparin-based anti-coagulation were eligible.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent before initiation of any study related procedures.
2. Be at least 18 years of age.
3. Patients requiring anticoagulation for the prophylaxis of thrombosis.
4. In the opinion of the Investigator, an alternative to heparin-based anticoagulant therapies is desirable.

Exclusion Criteria:

1. Confirmed pregnancy (if woman of child-bearing potential) (urine or serum pregnancy test).
2. Intracranial neoplasm, arteriovenous malformation or aneurysm.
3. Severe renal insufficiency (chronic or acute) with a GFR of < or equal to 30 mL/min as determined by measured or estimated creatinine clearance using Cockroft-Gault method or by estimated GFR using the MDRD formula.
4. Known allergy to desirudin or hirudin-derived drugs, or known sensitivity to any component of the product
5. Participation in other clinical research studies involving the evaluation of other investigational or FDA-approved drugs or devices within 30 days of enrollment (participation in observational studies of FDA-approved products is acceptable).
6. Refusal to undergo blood transfusion should it become necessary
7. Active bleeding or irreversible coagulation abnormality.
8. Uncontrolled hypertension defined as a blood pressure > or equal to 180/110 mmHg.
9. Patients requiring anticoagulation for left-ventricular assist device, intra-aortic balloon pump, veno-venous ultra filtration or ECMO.
10. Any other disease or condition which, in the judgment of the Investigator, would place a patient at undue risk by being enrolled in the trial, or cause inability to comply with the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 516 (Actual)
Dates: Start 2010-03; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dawn Bell, PharmD, Study Director — Canyon Pharmaceuticals, Inc.; Jerrold Levy, MD, FAHA, Principal Investigator — Emory University
Locations (15):
- United States (15):
  - University of Colorado Health Science Center, Aurora, Colorado
  - University of South Florida, Tampa General Hospital, Tampa, Florida
  - Saint Joseph's Research Institute, Atlanta, Georgia
  - Southeastern Center for Clinical Trials, Decatur, Georgia
  - Provena St. Joseph's Medical Center, Joliet, Illinois
  - Illinois Lung and Critical Care Institute, Peoria, Illinois
  - St. John's Mercy Medical Center, St Louis, Missouri
  - Overlook Hospital, Summit, New Jersey
  - Weill Cornell Medical College, New York, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - Forsyth Regional Medical Center, Winston-Salem, North Carolina
  - The Ohio State University Medical Center, Columbus, Ohio
  - Drexel University College of Medicine, Philadelphia, Pennsylvania
  - Research Concepts, Memorial Hermann Healthcare System, Houston, Texas
  - Carilion Roanoke Memorial Hospital, Roanoke, Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited between April 5, 2010 and February 18, 2011. Patients were recruited from inpatient medical and surgical services as well as surgical clinics when presenting for pre-operative services.
Period: Overall Study
Arm/Group | Desirudin
Started | 516
Completed | 516
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Desirudin
Number analyzed (Participants) | 516
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 387
  >=65 years | 129
Age Continuous [Mean (Standard Deviation); unit: years] | 59 (14.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 314
  Male | 202
Region of Enrollment [Number; unit: participants]
  United States | 516

OUTCOME MEASURES:

1. Primary Outcome: Major Bleeding
Description: Major bleeding is defined as clinically evident hemorrhage associated with a hemoglobin decrease ≥2 g/dL that leads to a transfusion of ≥2 units of whole blood or packed red cells outside of the peri-operative period (time from the start of the surgery or procedure and up to 12 hours after), or hemorrhage that is intracranial, retroperitoneal, or into a prosthetic joint.
Time Frame: 24 hours after last dose of study drug
Population: All patients receiving at least one dose of study drug
Measure: Number; unit: participants
Arm/Group | Desirudin
Number analyzed (Participants) | 516
participants | 0

2. Secondary Outcome: Thrombosis
Description: * New onset symptomatic thrombosis requiring medical or surgical intervention;
  * Death due to thrombosis defined as fatal pulmonary embolism, ischemic stroke, mesenteric thrombosis or myocardial infarction.
Time Frame: Up until 24 hours after last dose of study drug
Population: Patients who received at least one dose of study drug
Measure: Number; unit: participants
Arm/Group | Desirudin
Number analyzed (Participants) | 516
participants | 8

ADVERSE EVENTS:
Time Frame: up to 30 days after cessation of study drug
Arm/Group | Desirudin
Serious Adverse Events (participants affected / at risk) | 80/516
Other Adverse Events (participants affected / at risk) | 382/516
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Desirudin (N=516)
anemia (Blood and lymphatic system disorders) | 2 (2)
leukopenia (Blood and lymphatic system disorders) | 1 (1)
acute myocardial infarction (Cardiac disorders) | 4 (4)
atrial fibrillation (Cardiac disorders) | 5 (5)
cardiac failure congestive (Cardiac disorders) | 2 (2)
cardiogenic shock (Cardiac disorders) | 1 (1)
coronary artery disease (Cardiac disorders) | 1 (1)
abdominal distension (Gastrointestinal disorders) | 1 (1)
abdominal pain (Gastrointestinal disorders) | 2 (2)
colonic obstruction (Gastrointestinal disorders) | 1 (1)
constipation (Gastrointestinal disorders) | 3 (3)
gastric hemorrhage (Gastrointestinal disorders) | 4 (4)
gastrointestinal necrosis (Gastrointestinal disorders) | 1 (1)
hematemesis (Gastrointestinal disorders) | 1 (1)
ileus (Gastrointestinal disorders) | 1 (1)
nausea (Gastrointestinal disorders) | 2 (2)
pancreatic pseudocyst (Gastrointestinal disorders) | 1 (1)
rectal hemorrhage (Gastrointestinal disorders) | 1 (1)
small intestinal obstruction (Gastrointestinal disorders) | 7 (7)
vomiting (Gastrointestinal disorders) | 1 (1)
asthenia (General disorders) | 1 (1)
multi-organ failure (General disorders) | 2 (2)
cholecystitis acute (Hepatobiliary disorders) | 1 (1)
abdominal abscess (Infections and infestations) | 1 (1)
abdominal sepsis (Infections and infestations) | 1 (1)
bacterial infection (Infections and infestations) | 1 (1)
cellulitis (Infections and infestations) | 1 (1)
clostridium difficile colitis (Infections and infestations) | 2 (2)
diverticulitis (Infections and infestations) | 1 (1)
osteomyelitis (Infections and infestations) | 1 (1)
pelvic abscess (Infections and infestations) | 1 (1)
peridiverticular abscess (Infections and infestations) | 1 (1)
pneumonia (Infections and infestations) | 2 (2)
post-procedural infection (Infections and infestations) | 1 (1)
sepsis (Infections and infestations) | 3 (3)
septic shock (Infections and infestations) | 1 (1)
wound infection (Infections and infestations) | 1 (1)
gatrointestinal disorder postoperative (Injury, poisoning and procedural complications) | 1 (1)
gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 1 (1)
graft thrombosis (Injury, poisoning and procedural complications) | 1 (1)
postoperative ileus (Injury, poisoning and procedural complications) | 5 (5)
procedural nausea (Injury, poisoning and procedural complications) | 1 (1)
procedural pain (Injury, poisoning and procedural complications) | 1 (1)
procedural site reaction (Injury, poisoning and procedural complications) | 1 (1)
procedural vomiting (Injury, poisoning and procedural complications) | 1 (1)
splenic hematoma (Injury, poisoning and procedural complications) | 1 (1)
subdural hematoma (Injury, poisoning and procedural complications) | 1 (1)
white blood cell count increased (Investigations) | 1 (1)
dehydration (Metabolism and nutrition disorders) | 1 (1)
failure to thrive (Metabolism and nutrition disorders) | 1 (1)
pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
embolic stroke (Nervous system disorders) | 1 (1)
syncope (Nervous system disorders) | 3 (3)
hydronephrosis (Renal and urinary disorders) | 1 (1)
renal failure (Renal and urinary disorders) | 3 (3)
renal failure acute (Renal and urinary disorders) | 5 (5)
uretic obstruction (Renal and urinary disorders) | 1 (1)
pelvic fluid collection (Reproductive system and breast disorders) | 1 (1)
pelvic pain (Reproductive system and breast disorders) | 1 (1)
vaginal hemorrhage (Reproductive system and breast disorders) | 1 (1)
atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
bronchial secretion retention (Respiratory, thoracic and mediastinal disorders) | 1 (1)
chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
diaphragmatic hernia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 (4)
pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 (4)
cholecystectomy (Surgical and medical procedures) | 1 (1)
deep vein thrombosis (Vascular disorders) | 3 (3)
haematoma (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Desirudin (N=516)
constipation (Gastrointestinal disorders) | 76 (76)
nausea (Gastrointestinal disorders) | 76 (76)
procedural pain (Injury, poisoning and procedural complications) | 59 (59)
anemia (Blood and lymphatic system disorders) | 45 (45)
breath sounds abnormal (Respiratory, thoracic and mediastinal disorders) | 41 (41)
pyrexia (General disorders) | 39 (39)
hypophosphataemia (Metabolism and nutrition disorders) | 38 (38)
tachycardia (Cardiac disorders) | 37 (37)
asthenia (General disorders) | 36 (36)
anemia postoperative (Injury, poisoning and procedural complications) | 33 (33)
oxygen saturation decrease (Respiratory, thoracic and mediastinal disorders) | 32 (32)
oedema peripheral (Vascular disorders) | 31 (31)
vomiting (Gastrointestinal disorders) | 31 (31)
hyperglycemia (Metabolism and nutrition disorders) | 30 (30)
hypokalemia (Metabolism and nutrition disorders) | 27 (27)
hypotension (Cardiac disorders) | 27 (27)
generalised oedema (General disorders) | 26 (26)
hypocalcemia (Metabolism and nutrition disorders) | 26 (26)

LIMITATIONS AND CAVEATS:
This was a multi-center, single-arm, observational safety trial. The lack of an active comparator does not allow us to make conclusions about the relative safety and efficacy of the product.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less